CLINICAL TRIAL: NCT03794934
Title: Development and Efficacy of Individualized Professional Education Based on New Glucose Management Devices in Patients With Type 1 Diabetes Mellitus
Brief Title: Structured Education Based on New Glucose Management Devices in Patients With Type 1 Diabetes Mellitus
Acronym: Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jae Hyeon Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-12-108
Record Dates: First submitted 2019-01-04; First posted 2019-01-07 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Continuous Glucose Monitoring; Insulin pump; Structured Education
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: CGM apply followed by structured education of CGM
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Without structured education when applying CGM for 3months, and as a sequential extension clinical trial, after 3 months, structured education is provided, followed by CGM apply
  Interventions: Behavioral: Structured Education for new glucose management devices
- Intervention (Active Comparator): provide structured education when applying CGM for 3 months
  Interventions: Behavioral: Structured Education for new glucose management devices

INTERVENTIONS:
Behavioral: Structured Education for new glucose management devices — Individualized professional education based on new glucose management devices in patients with type 1 diabetes mellitus

SUMMARY:
Continuous glucose monitoring (CGM) and insulin pump, a new medical device, have been proved and highly recommended in the treatment of type 1 diabetes patients worldwide, and related technology development and market are growing rapidly.

In order to maximize the medical and socioeconomic effects of the latest blood glucose devices including CGM and insulin pump, structured education is necessary. In this study, we will develop patient-oriented structured education for patients with type 1 diabetes mellitus when applying CGM, and we will assess the efficacy of this education protocol for patients with type 1 diabetes using CGM.

DETAILED DESCRIPTION:
In 50 patients with type 1 diabetes with over 7% of glycated hemoglobin, whose blood glucose level is not well controlled, and who are undergoing multiple daily insulin injection therapy or insulin pump therapy, continuous glucose monitoring (CGM) is applied to obtain basal continuous glucose levels for 1 week (window period of 2 week).

These 50 patients are 1:1 randomly assigned to 2 groups including control group and intervention group. Control group (n=25) applied CGM without structured education and after 3 months of applying CGM, continuous glucose data for 2 consecutive weeks and HbA1c level, and other glycometabolic parameters are collected. As a sequential extension clinical trial, those 25 patients in control group are provided structured education, followed by applying CGM for 3 months. Continuous glucose levels for 2 consecutive weeks and HbA1c level, and other glycometabolic parameters are collected.

In Intervention group (n=25), structured education program is provided for each patient from the time of enrollment, followed by applying CGM for 3 months. Continuous glucose levels for 2 consecutive weeks and HbA1c level and other blood tests are performed after the 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old - under 70 years old patients with Type 1 diabetes
* Those who plan to use CGM G5
* Patients who consented to use CGM G5 in conjunction with Clarity
* Those who are using multiple insulin injections or insulin pumps for at least 3 months
* Those whose fasting c-peptide <0.6 ng / dL, or stimulated c-peptide <1.8 ng / dL
* Those with a glycated hemoglobin of 7.0% or more within the last 3 months
* Those who have never used a CGM for more than a month
* For women of childbearing age, those who agree to use appropriate contraception during the trial
* Those who voluntarily signed the agreement after the explanation of the clinical trial

Exclusion Criteria:

* Those with a history of severe hypoglycemia and acute ketoacidosis within the last 3 months
* Patients with chronic renal function greater than or equal to stage 4 (estimated glomerular filtration rate [assessed by MDRD (modification of diet in renal disease] <30 )
* Patients with acute myocardial infarction, unstable angina, coronary artery disease or stroke within the last 3 months
* Patients with adrenal insufficiency, pituitary dysfunction, medically uncontrolled hyperthyroidism or hypothyroidism
* Those taking medications that can affect the glucose metabolism (eg, corticosteroids, immunostimulants, etc.)
* Pregnant and lactating women
* A person who is deemed unsuitable for participation in clinical trials by examiners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in target range 70-180 mg/dL | 3months (control and intervention groups) and 6months (for extension study in control group)
  Percentage of time in target range 70-180 mg/dL by continuous glucose monitoring system

SECONDARY OUTCOMES:
Percentage of time in level 2 hypoglycemia (<54mg/dL) | 3months (control and intervention groups) and 6months (for extension study in control group)
  Percentage of time in level 2 hypoglycemia (<54mg/dL) by continuous glucose monitoring system
Percentage of time in level 1 hypoglycemia (<70-54mg/dL) | 3months (control and intervention groups) and 6months (for extension study in control group)
  Percentage of time in level 1 hypoglycemia (<70-54mg/dL) by continuous glucose monitoring system
Percentage of time in level 1 hyperglycemia (>180mg/dL) | 3months (control and intervention groups) and 6months (for extension study in control group)
  Percentage of time in level 1 hyperglycemia (>180mg/dL) by continuous glucose monitoring system
Percentage of time in level 2 hyperglycemia (>250mg/dL) | 3months (control and intervention groups) and 6months (for extension study in control group)
  Percentage of time in level 2 hyperglycemia (>250mg/dL) by continuous glucose monitoring system
Glycemic variability, reported as coefficient of variance (CV) | 3months (control and intervention groups) and 6months (for extension study in control group)
  Glycemic variability, reported as coefficient of variance (CV) by continuous glucose monitoring system
Glycemic variability, reported as standard deviation (SD) | 3months (control and intervention groups) and 6months (for extension study in control group)
  Glycemic variability, reported as standard deviation (SD) by continuous glucose monitoring system
Mean glucose by continuous glucose monitoring system | 3months (control and intervention groups) and 6months (for extension study in control group)
  Mean glucose by continuous glucose monitoring system
HbA1C | 3months (control and intervention groups) and 6months (for extension study in control group)
  HbA1C
glycated albumin | 3months (control and intervention groups) and 6months (for extension study in control group)
  glycated albumin
Personalized education time for each patient | baseline (intervention group) and 3months (for extension study in control group)
  Personalized education time for each patient
Frequency of hypoglycemia | 3months (control and intervention groups) and 6months (for extension study in control group)
  Frequency of hypoglycemia
Adverse event | 3months (control and intervention groups) and 6months (for extension study in control group)
  Adverse event occurred
Percentage of time in target range 70-180 mg/dL | 6months (for extension study in control group)
  Percentage of time in target range 70-180 mg/dL by continuous glucose monitoring system

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoo JH, Kim G, Lee HJ, Sim KH, Jin SM, Kim JH. Effect of structured individualized education on continuous glucose monitoring use in poorly controlled patients with type 1 diabetes: A randomized controlled trial. Diabetes Res Clin Pract. 2022 Feb;184:109209. doi: 10.1016/j.diabres.2022.109209. Epub 2022 Jan 19. PMID 35065101